CLINICAL TRIAL: NCT06859697
Title: The Efficacy and Safety of Herbal Medicine Treatment for Obese Patients With Spinal and Joint Pain: A Pragmatic Randomized Controlled Pilot Clinical Trial
Brief Title: The Efficacy and Safety of Herbal Medicine Treatment for Obese Patients With Spinal and Joint Pain
Acronym: Obesity PCT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JS-CT-2025-03; Jaseng Medical Foundation (Other: Jaseng Medical Foundation)
Record Dates: First submitted 2025-02-26; First posted 2025-03-05 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Obesity and Overweight
Keywords: Obesity Herbal Medicine
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Herbal Medicine Group (Experimental): Participants in the herbal medicine treatment group will visit the clinic every 14 days for prescription and follow-up observations. Herbal medicine will be prescribed in 14-day doses, and participants will orally take a total of 42 days' worth of herbal medicine during the treatment period.
  This study is a pragmatic clinical trial, and there are no restrictions on the types of herbal medicine used. Prescriptions will be made at the discretion of the medical staff, with the primary goal of improving obesity.
  All prescriptions will be made by Korean medicine doctors with at least five years of clinical experience.
  After the prescription is issued, the herbal medicine will be delivered to participants via courier for consumption. Participants will be instructed to store all herbal medicine in a refrigerator.
  Compliance with herbal medicine consumption will be confirmed by counting the remaining doses during participants' visits and recording the results.
  Interventions: Procedure: Herbal medicine treatment
- Life Guidance Group (Active Comparator): Educational materials will be distributed, and education sessions will be conducted.
  Interventions: Procedure: Life Guidance

INTERVENTIONS:
Procedure: Herbal medicine treatment — Herbal medicine treatment is a treatment using complex extract of medicinal herbs prescribed by a Korean medicine doctor who has completed specialized education to diagnose the health condition and symptoms of patients
  Arms: Herbal Medicine Group
Procedure: Life Guidance — Educational materials will be distributed, and education on daily life management for weight loss will be conducted. The educational materials consist of information on the definition and causes of obesity, explanations on weight reduction and daily life management applicable to various situations such as exercise and diet, and the effects of these practices.
  Arms: Life Guidance Group

SUMMARY:
This study is a pragmatic pilot randomized controlled trial aimed at investigating the effectiveness of herbal medicine treatment for obese patients with spinal and joint pain, using a control group receiving lifestyle guidance.

DETAILED DESCRIPTION:
0. Background Obesity has been defined as a chronic disease requiring long-term treatment by the World Health Organization (WHO). Additionally, an increase in body fat is associated with a higher prevalence of musculoskeletal pain and related disorders. Therefore, this study aims to evaluate the efficacy of herbal medicine treatment by investigating whether a reduction in obesity affects spinal and joint pain in obese patients, who constitute a significant proportion of patients visiting Korean medicine clinics and hospitals for spinal and joint pain.

1. Patient Recruitment and Screening Phase

1. Patient Recruitment Forty patients meeting the inclusion/exclusion criteria will be recruited starting from the date of IRB registration. Researchers will use block randomization to allocate participants. After obtaining written consent from patients who meet the criteria, they will be assigned to the study. The probability of assignment to each group will be 1:1.
2. Allocation Concealment and Blinding Since blinding is not feasible for this study, it will be conducted as an open-label clinical trial. However, assessor blinding will be implemented. The evaluator, who will not participate in the intervention and will be blinded to group allocation, will conduct assessments in a separate space before the intervention. This role will be performed by a research nurse or a specialist in training.

2. Treatment and Evaluation Phase

1. Control and Experimental Groups The experimental group will receive herbal medicine treatment in addition to standard care, while the control group will receive lifestyle guidance only. Both groups will be provided with identical educational materials and guidance on lifestyle modifications aimed at weight loss.

   The educational materials will include information on the definition and causes of obesity, as well as explanations on weight reduction and lifestyle management applicable to various situations, including diet and exercise.

   Lifestyle guidance will be based on the provided materials. During the first visit, participants will receive comprehensive education on the study materials. Follow-up education sessions will be conducted every two weeks for a total of six weeks, during which changes in participants' symptoms will also be evaluated.

   Both groups will receive lifestyle education under identical conditions to evaluate the additional effects of herbal medicine treatment.
2. Study Duration and Observation Points The total participation period for each subject will be 12 weeks, including a 6-week treatment period and a 6-week follow-up period.

   Baseline data will be collected at the time of study enrollment (Week 0), and the primary endpoint will be at Week 6.

   Data will be collected during visits at Week 0, Week 2, and Week 4 during the treatment period, as well as during follow-up visits at Week 6 (primary endpoint), Week 8, and Week 12.
3. Data Collection for Evaluation i. Primary Outcome The primary outcome will be the BMI at Week 6, after the completion of the treatment intervention.

ii. Secondary Outcomes

Secondary outcomes will be assessed at Week 0, Week 2, Week 4, Week 6 (primary endpoint), Week 8, and Week 12. The following indicators will be evaluated:

Body fat percentage Body fat mass Skeletal muscle mass Body weight Visceral fat level Quality of life (EQ-5D-5L) IWQOL-Lite (Impact of Weight on Quality of Life - Lite) The most painful area in the spinal and joint regions NRS (Numeric Rating Scale) for pain intensity Adherence to the intervention Adverse effects

3. Follow-Up Phase After the 6-week intervention period, a 6-week follow-up will be conducted to assess changes in the participants' symptoms.

At Weeks 6, 8, and 12, evaluations will be conducted using the same parameters as during the treatment visits, including the primary outcome (BMI) and secondary outcomes (body weight, body fat percentage, body fat mass, skeletal muscle mass, EQ-5D, IWQOL-Lite, the most painful spinal/joint area, pain intensity at that site, adherence, and adverse effects). The time window for follow-up evaluations will be ±5 days for Week 6 and ±7 days for Weeks 8 and 12.

Blood tests will be conducted at Week 6, aligned with the start of herbal medicine treatment. The blood test parameters will be the same as those performed during the screening phase.

4. Monitoring

Although this is a researcher-initiated clinical study, monitoring will be conducted by a third party in accordance with the institution's HRPP (Human Research Protection Program) policy and KCGP (Korean Good Clinical Practice) guidelines. The purpose of monitoring is to ensure that the following are maintained throughout the study period and to prevent recurrence of any non-compliance through proper reporting procedures:

Monitoring intervals will be appropriately spaced, and the frequency will depend on the rate of participant enrollment and the data collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 19 years or older but under 70 years.
* Individuals with a BMI of 25 kg/m² or higher, meeting the Asia-Pacific obesity criteria.
* Individuals experiencing spinal or joint pain, with the most severe pain rated as NRS 5 or higher.
* Individuals who voluntarily agree to participate in the clinical trial and sign the consent form.

Exclusion Criteria:

* Presence of findings on X-ray examination of the pain site, such as acute fractures or dislocations, requiring surgical intervention.
* Diagnosis of specific diseases that may cause secondary obesity (e.g., Cushing's syndrome, hypothyroidism, insulinoma, adult growth hormone deficiency, etc.).
* Current use of medications related to obesity treatment or a history of taking such medications within the past month.
* Presence of other chronic diseases that may interfere with treatment efficacy or interpretation of results, such as stroke, myocardial infarction, kidney disease, active hepatitis, diabetic neuropathy, dementia, epilepsy, etc.
* Current use of steroids, immunosuppressants, psychiatric medications, or other drugs that may affect study outcomes.
* Unsuitability or safety concerns for herbal medicine treatment: individuals with conditions or post-surgical complications affecting drug absorption or digestion, severe liver disease, or kidney disease.
* Pregnant or planning to become pregnant, or currently breastfeeding.
* Participation in other clinical trials, except for observational studies without therapeutic intervention.
* Difficulty in providing informed consent.
* Other cases where the investigator deems participation in the clinical study inappropriate.

Ages: 19 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
BMI(Body Mass Index) | Change from baseline to Week 6
  Body weight (kg) divided by the square of height (m) is used as a diagnostic criterion for obesity. Based on the significant increase in obesity-related diseases associated with body mass index (BMI), the Asia-Pacific region and the Korean Society for the Study of Obesity have established the criteria as follows: a BMI of 23 kg/m² or higher is classified as overweight or pre-obesity, and a BMI of 25 kg/m² or higher is classified as obesity.

SECONDARY OUTCOMES:
Body Fat Percentage | Baseline(Week 0), Week 2, Week 4, Week 6, Week 8, Week 12
  Body fat percentage (percent body fat, PBF, %fat) is the proportion of body fat relative to total body weight. Obesity classification based on body fat percentage is as follows: for men, less than 10.0% is classified as underweight, 10.0-20.0% as normal, 20.0-25.0% as overweight, and 25.0% or higher as obesity; for women, less than 18.0% is classified as underweight, 18.0-28.0% as normal, 28.0-33.0% as overweight, and 33.0% or higher as obesity.
Body fat mass | Baseline(Week 0), Week 2, Week 4, Week 6, Week 8, Week 12
  Body fat mass refers to the absolute amount of fat in the body, measured in kilograms (kg). It represents the total weight of fat tissue in the body and is an important indicator for assessing obesity and overall body composition. Unlike body fat percentage, which is a relative measure, body fat mass provides an absolute value, making it useful for tracking changes in fat levels over time, especially during weight management or fitness programs.
Skeletal Muscle Mass | Baseline(Week 0), Week 2, Week 4, Week 6, Week 8, Week 12
  Skeletal muscle mass refers to the total weight of skeletal muscles in the body, typically measured in kilograms (kg). Skeletal muscles are responsible for voluntary movements and play a crucial role in physical activity, metabolism, and overall health. This measurement is used to assess muscle development and monitor changes due to exercise, aging, or medical conditions
Body weight | Baseline(Week 0), Week 2, Week 4, Week 6, Week 8, Week 12
  Body weight refers to the total mass of an individual's body, typically measured in kilograms (kg) or pounds (lbs). It includes the combined weight of bones, muscles, fat, organs, fluids, and other tissues. Body weight is a fundamental parameter for assessing overall health and is often used in conjunction with other measurements, such as body fat percentage, skeletal muscle mass, and BMI, to evaluate physical fitness, nutritional status, and the risk of developing obesity-related diseases.
Visceral fat level | Baseline(Week 0), Week 2, Week 4, Week 6, Week 8, Week 12
  Visceral fat level refers to the amount of fat stored around internal organs in the abdominal cavity, such as the liver, pancreas, and intestines. In InBody devices, visceral fat level is expressed on a scale ranging from 1 to 20, where a level below 10 is generally considered healthy, while a level of 10 or higher indicates excessive visceral fat that may require management.
5-Level EuroQol-5 Dimension (EQ-5D-5L) | Baseline(Week 0), Week 2, Week 4, Week 6, Week 8, Week 12
  The 5-Level EuroQol-5 Dimension (EQ-5D-5L) is one of the most widely used indirect measurement methods for calculating the quality weight of a specific health state. It evaluates health status from multiple perspectives and utilizes pre-assigned preference scores for each functional level to indirectly calculate the quality weight of a particular health condition. The EQ-5D-5L consists of five items, each addressing the degree of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each item is assigned a specific weight based on its level, and a preference score calculation formula is provided using these weights and constants.
IWQOL-Lite (Impact of Weight on Quality of Life - Lite) | Baseline(Week 0), Week 2, Week 4, Week 6, Week 8, Week 12
  The IWQOL-Lite is a questionnaire tool developed to assess the impact of weight on quality of life and is primarily used in obesity research and evaluating the effectiveness of weight loss treatments. It is a simplified version of the IWQOL (Impact of Weight on Quality of Life) and consists of 31 items. The questionnaire is divided into five subscales: physical function, self-esteem, sexual life, interpersonal stress, and work-related activities.
Areas of Spinal and Joint Pain | Baseline(Week 0), Week 2, Week 4, Week 6, Week 8, Week 12
  To investigate the primary pain areas in the spinal and joint regions of obese patients, the severity of pain in the single most painful area is assessed.
NRS (Numeric Rating Scale) | Baseline(Week 0), Week 2, Week 4, Week 6, Week 8, Week 12
  The Numeric Rating Scale (NRS) is used to assess the severity of pain in the single most painful area. Patients rate their pain on a scale from 0 to 10, where 0 represents "no pain at all" and 10 represents "the worst pain imaginable or unbearable pain." This scale provides a simple and effective way to quantify pain levels for clinical evaluation and treatment planning.
Adherence | Week 2, Week 4, Week 6
  To evaluate treatment adherence, for participants in the herbal medicine treatment group, the total number of prescribed herbal medicine packs and the number of consumed packs are assessed from Week 0 to Week 6 and recorded in the Case Report Form (CRF).
  Additionally, for all participants, the number of days they adhered to dietary and exercise regimens is also investigated and documented in the CRF. This comprehensive adherence evaluation helps ensure accurate monitoring of participants' compliance with treatment protocols and lifestyle modifications.

OTHER OUTCOMES:
Adverse Event (AE) | Week 2, Week 4, Week 6, Week 8, Week 12
  An adverse event refers to any undesirable and unintended objective sign, subjective symptom, or disease that occurs after a clinical trial procedure, and it does not necessarily have to have a causal relationship with the procedure. During the study period, adverse events are collected through participants' symptom reports and researchers' observations, and the type of adverse event along with its causal relationship to the intervention is recorded in the Electronic Medical Record (EMR). In case of an adverse event, follow-up monitoring is conducted, and any severe adverse event is promptly reported. The causality of adverse events is classified into six levels based on the WHO-UMC causality categories: Certain (1), Probable/Likely (2), Possible (3), Unlikely (4), Conditional/Unclassified (5), and Unassessable/Unclassifiable (6). The severity of adverse events is assessed using the Spilker classification, dividing them into three levels: Mild (1), which does not re

CONTACTS AND LOCATIONS:
Overall Officials: In-Hyuk Ha, PhD, Principal Investigator — Jaseng Medical Foundation
Locations (1):
- Jaseng Hospital of Korean Medicine, Seoul, Gangnam-Gu, South Korea

IPD SHARING:
Plan to Share IPD: No